CLINICAL TRIAL: NCT06292247
Title: Effectiveness of Cognitive Behavioral Therapy and Auricular Plaster Therapy on Managing Child Anxiety in Dental Office
Brief Title: Effectiveness of CBT and APT on Managing Child Anxiety in Dental Office
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Reina Abed, Principle Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A0503023
Record Dates: First submitted 2024-02-13; First posted 2024-03-05 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Dental Anxiety
Keywords: dental anxiety (DA); Cognitive behavioral therapy (CBT); Auricular Plaster Therapy (APT); Tell Show Do (TSD)
MeSH Terms: interventions — Cognitive Behavioral Therapy; Acupressure

STUDY DESIGN:
Intervention Model Description: Group 1 (CBT) Group 2 (APT) Group3 (control TSD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive behavioral therapy group (Experimental): CBT is based on the principle that, the way we think profoundly impacts the way we feel and behave. Therefore, learning to think differently can enable the child to feel and act differently. It is a multi-component therapy that companies cognitive (cognitive restructuring) and behavioral (relaxation and distraction) interventions to change these maladaptive cognitions, which change the emotional distress and problematic behaviors. The following techniques were used in our research in a row, unrelated play, animated video modeling, stress-ball relaxation technique, audio music therapy, and positive reinforcement. These have been used effectively to manage children's anxiety during the dental appointment.
  Interventions: Behavioral: Auricular plaster therapy; Behavioral: Tell Show Do
- Auricular Plaster Therapy group (Experimental): APT intervention involves the application of plaster with seeds on specific points of the outer ear, known as auricular points (acupoints). According to Traditional Chinese Medicine, these points correspond to various regions of the body. Applying pressure to these points (acupressure) will stimulate and regulate energy flow throughout the body. This process is believed to restore balance and harmony within the body's system and achieve a therapeutic effect e.g. (anxiety reduction)
  Interventions: Behavioral: Cognitive behavioral therapy; Behavioral: Tell Show Do
- Control group (Tell show do) (Experimental): TSD is considered the cornerstone of behavior management techniques. It aims to introduce the child to the dental setting before commencing any procedure. With the TSD technique, the child should be informed about the process with a demonstration of the dental procedure using a simulator.
  Interventions: Behavioral: Cognitive behavioral therapy; Behavioral: Auricular plaster therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — CBT aims to treat anxiety by restructuring unfavorable beliefs and controlling negative thoughts so as to reduce dental anxiety.
  Arms: Auricular Plaster Therapy group; Control group (Tell show do)
Behavioral: Auricular plaster therapy — APT involves the application of plaster with seeds on specific points of the outer ear, known as auricular points (acupoints). This process is believed to restore balance and harmony within the body's system and achieve a therapeutic effect (e.g. reduce anxiety)
  Other Names: acupressure
  Arms: Cognitive behavioral therapy group; Control group (Tell show do)
Behavioral: Tell Show Do — TSD is composed of 3 phases. The Tell phase involves an age-appropriate explanation of the procedure. The Show phase is used to demonstrate a procedure up to the point where the instrument is performed. The Do phase is then initiated, and the treatment is performed.
  Other Names: TSD
  Arms: Auricular Plaster Therapy group; Cognitive behavioral therapy group

SUMMARY:
This study was conducted to the Effectiveness of Cognitive Behavioral Therapy and Auricular Plaster Therapy on Managing Child Anxiety in Dental Office.

DETAILED DESCRIPTION:
This study is to:

1. Assess and compare the effect of cognitive behavioral therapy and auricular plaster therapy on children's anxiety in dental situations.
2. Improve child behavior and cooperation and evaluate the parental acceptance of these behavioral management techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children (4-7) years old, without systemic, congenital, or mental disorders nor deformities affecting the external auditory meatus.
2. Presence of dental anxiety.
3. Not requiring urgent dental treatment, with the presence of a Class I carious lesion on one of the primary molars.
4. No previous application of the guided CBT.

Exclusion Criteria:

1. Refusal to participate by either the children or their parents/guardians
2. Previous receiving acupuncture and moxibustion therapy.
3. Children who had taken sedative drugs at the time of the appointment.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Venham Clinical Anxiety Scale | Up to 12 weeks
  Observational anxiety scale, by choosing a number from 0 to 5 as claimed by the scales at specific time spots of the dental visit. The higher the score, the greater the level of anxiety and the poorer the cooperation of a child
Heart Rate to detect the anxiety. | Up to 12 weeks
  It is a biological parameter and the elevation of pulse rate is an indicator for anxiety
RMS-Self Pictorial scale to detect the anxiety. | Up to 12 weeks
  It is a self-report scale, ranging from (1 to 5). The scale was scored by giving a value of one to very happy and five to very unhappy face. (A higher score indicates more anxiety)

SECONDARY OUTCOMES:
Parental acceptance of the behavior management technique | Up to 12 weeks
  The parental acceptance rating will be determined on a five-point Likert-type scale ranging from 1 (highly acceptable) to 5 (highly unacceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Reina N Abed, Master, Principal Investigator — Mansoura University; Salwa M Awad, Prof, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University; Ahmad H Wahba, PhD, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University
Locations (1):
- Faculty of dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol to other researchers
Supporting Information: Study Protocol
Time Frame: Within 6 months
Access Criteria: For anyone